CLINICAL TRIAL: NCT06102538
Title: "Hachi Barie" Project - A Multidisciplinary Program to Accompany Severely Obese Teenagers in the Weight Loss Process for the Benefit of Their Recruitment Into the Israel Defense Forces
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Orit Hamiel, Head of pediatric endocrinology and diabetes unit, Sheba Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0392-23-SMC
Record Dates: First submitted 2023-10-09; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Morbid Obesity
Keywords: morbid obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Intervention Model Description: The structure of the meetings - once a week
  1. An hour and a half of physical activity adapted to the ability of teenagers with morbid obesity.
  2. An hour and a half of training and education, which will include:
     * 10 group sessions with a dietician 45 minutes each session
     * 10 group meetings with a mental health staff member, 45 minutes per meeting (at least two of the meetings will be designated for a joint cooking workshop with the parents)
     * 6 meetings with IDF personnel, value meetings: the structure of the army, integration into the army, etc.
  3. Meetings for parents - will include guidance from a nutritionist, exercise for parents, resilience for parents.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morbid obese adolescents with comorbidity (Active Comparator): A weekly intervention of physical education, group psychological support, and nutrition education.
  Interventions: Behavioral: # The importance of service in the IDF # Physical activity # Healthy nutrition # Psychological support
- Obese children who do not participate in this intervention (No Intervention): This group of adolescents will continue the routine treatment in the clinic

INTERVENTIONS:
Behavioral: # The importance of service in the IDF # Physical activity # Healthy nutrition # Psychological support — # Education for the importance of service in the IDF # Education and training for physical activity adapted to abilities # Training for a healthy diet # Psychological support
  Arms: Morbid obese adolescents with comorbidity

SUMMARY:
Teenagers with body mass values (BMI) above 35 kg/m2 and co-morbidity are designated for medical disqualification from service in the IDF. Data show that there has been an increase in the incidence of these teenagers, specifically among the lower socioeconomic status. The purpose of this pilot study is to carry out an intervention Based lifestyle modification among a group of boys and girls with morbid obesity accompanied by a comorbidity that disqualifies them from service in the IDF.

Definition of success: meeting the threshold of weight and health status that allows recruitment into the IDF.

Criteria for finding candidates:

* Boys and girls from the age of 15 who suffer from morbid obesity and comorbidity that may prevent their enlistment in the IDF. (This age range was chosen to allow an ideal period of at least one year to make a significant change).
* Boys and girls who have their own and their family's willingness and commitment to participate in the process
* A basic state of health that allows participation in the program. The screening process will be done by the staff of the endocrine unit, under the management of Prof. Orit Pinhas-Hamiel.

Duration of intervention:

26 weekly sessions for the trainees. The duration of the meeting will be about three hours in the afternoon A decision whether to extend the duration of the intervention will be taken according to the initial results of the program.

Activity location:

Potential sites vary: Sheba// academic complex // military base for trainees. Number of participants - 25, (dropout expected 30%) Research goals (main content elements in the program) - there are 3 main content areas (of similar importance)

* Education about the importance of service in the IDF and the opportunities inherent in it
* Ability-adapted physical activity education and training
* Guidance for a healthy diet
* Psychological support [The medical accompaniment to the program will take place on the basis of the patients' mother clinics and the medical follow-up of them will be done separately].

DETAILED DESCRIPTION:
The purpose of the program:

* Readiness for recruitment into the IDF, both in terms of recruitment criteria, and in terms of motivation
* Candidates: teenagers aged 15 and over, who, based on their weight and associated morbidity, can be assumed to be exempt from conscription. Boys and girls motivated for change.

Half-yearly program (26 sessions) with an option to extend.

* The location of the activity. Closed meetings at the college in Kiryat Ono, meetings will also be planned at the Wingit Institute, and at the IDF base (if possible).
* Number of participants for the initial pilot about 25 participants. More groups will be opened later.
* Before the start, the candidates will be screened by psychologists from the pediatric endocrinology unit,
* Before the start, the candidates will undergo a comprehensive medical examination by a pediatrician and endocrinologist, which will include height, weight, blood pressure test, waist circumference, Bio-Impedence
* In the first and last meeting, the physical ability will be assessed by me

  1. 6-minute walk test (6MWT)
  2. Balance tests
* Dynamic balance test - star excursion balance test
* Stork Balance Stand Test, time measurement. 3. Muscle strength tests: pressing force with a hand dynamometer. Questionnaires
* In the first and last meeting the participants will fill
* Questionnaires of eating habits FFQ, as well as pickiness in food
* Questionnaires about motivation, self-efficacy, depression

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls ages 15 -19 years
* Obesity - BMI >30-40 Kg/m2
* Additional morbidity ( Type 2 diabetes, Hypertension)
* A basic state of health that allows participation in the program.
* Boys and girls who have their own and their family's willingness and commitment to participate in the process
* Expected to be exempt from enlistment in the IDF

Exclusion Criteria:

* retardation
* a syndrome that does not allow integration into the group
* significant morbidity that prevents physical activity according to the decision of the attending physician.

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-10-10 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Weight loss | 1 year
  The change in weight from the baseline of the study to the end of the study
Psychological well-being - improvement in coherence | 3 and 6 months
  Sense of Coherence Scale - by Antonovsky

SECONDARY OUTCOMES:
Improving eating habits | 3 and 6 months
  Eating habits Food frequency Questionnaire (FFQ) A screening questionnaire adapted to Israel for food consumption according to the principles of the Mediterranean diet -I-MEDAS Israeli MABAT Questionnaire - Israeli Ministry of Health
Improvement in physical fitness | 3 and 6 months
  Improvement in physical fitness
  The 6-minute walking test (6MWT) - an acceptable walking test
An increase in motivation for the IDF recruitment process | 3 and 6 months
  Number of participant who will eventually be recruited to the army
Decrease in Depression | 3 and 6 months
  A decrease in the level of depression - Using PHQ9-
Increase in social support | 3 and 6 months
  Scale of Perceiver Social Support MSPSS by (Ziment, Dahlem, Ziment and Fanley, 1988)
Improvement in quality of life | 3 and 6 months
  Improvement in quality of life -Improvement in quality of life - (IWQOL-Kids)
Improvement in self-efficacy - | 3 and 6 months
  Self Efficacy questionnaire by Chen, Gully and Eden 2001
Balance test: testing balance | 3 and 6 months
  Dynamic balance test - Star Excursion Balance Test
Balance test: testing balance time measurement. | 3 and 6 months
  Stork Balance Stand Test

CONTACTS AND LOCATIONS:
Locations (1):
- Endocrine and Diabetes Unit, Sheba Medical Center, Ramat Gan, Israel